CLINICAL TRIAL: NCT01459809
Title: A Multinational, Open Label, Randomized, Active-controlled, 3-arm Parallel Group, 24-week Study Comparing the Combination of Glimepiride and Metformin Versus Glimepiride and Metformin Alone in Patients With Type 2 Diabetes
Brief Title: Efficacy and Safety Comparison of Metformin/Glimepiride Combination Versus Each Compound Alone in New Diagnosed Type 2 Diabetes Patients
Acronym: RECOMMEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLIME_R_05809; U1111-1119-9984 (Other: UTN)
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM 1: glimepiride alone (Experimental): 24-week treatment period: After randomization, starting dose will be of 2 mg /day or 1 mg/day of glimepiride if Fasting Plasma Glucose (FPG) at baseline < 180 mg/dL (10 mmol/L) taken once in the morning before breakfast. The treatment's dose will be increased every 2 weeks up to the maximum tolerated dose of 4 mg, and adjusted throughout the 24-week treatment period according to fasting Self Monitored Plasma Glucose (SMPG) values in the objective to obtain fasting SMPG values ≤ 130mg/dL (7.2mmol/L) and > 70 mg/dL (3.9mmol/L) without symptomatic hypoglycemia.
  Interventions: Drug: GLIMEPIRIDE
- ARM 2: metformin alone (Experimental): 24-week treatment period: After randomization, starting dose will be of 500 mg of metformin twice a day during or after meals. The treatment's dose will be increased every 2 weeks up to the maximum tolerated dose of 2000 mg, and adjusted throughout the 24-week treatment period according to fasting SMPG values in the objective to obtain fasting SMPG values ≤ 130mg/dL (7.2mmol/L) and > 70 mg/dL (3.9mmol/L) without symptomatic hypoglycemia.
  Interventions: Drug: METFORMIN
- ARM3: Glimepiride/metformin free combination (Experimental): 24-week treatment period: After randomization, starting dose will be of 2 mg /day or 1 mg/day of glimepiride if FPG at baseline < 180 mg/dL (10 mmol/L) taken once in the morning and 500 mg of metformin twice a day taken during or after meals. The treatment's dose will be increased every 2 weeks up to the maximum tolerated dose of 4 mg of glimepiride and 2000 mg of metformin, and adjusted throughout the 24-week treatment period according to fasting SMPG values in the objective to obtain values ≤.
  Interventions: Drug: GLIMEPIRIDE; Drug: METFORMIN

INTERVENTIONS:
Drug: GLIMEPIRIDE — Pharmaceutical form: oral
  Route of administration: oral
  Other Names: HOE490
  Arms: ARM 1: glimepiride alone; ARM3: Glimepiride/metformin free combination
Drug: METFORMIN — Pharmaceutical form: oral
  Route of administration: oral
  Arms: ARM 2: metformin alone; ARM3: Glimepiride/metformin free combination

SUMMARY:
Primary Objective:

- To demonstrate the superiority of glimepiride and metformin free combination in comparison to glimepiride or metformin alone in terms of Hb1Ac reduction during a 24-week treatment period in patients with type 2 diabetes mellitus.

Secondary Objectives:

- To assess the effects of the free combination of glimepiride and metformin in comparison to glimepiride or metformin alone on:

* Percentage of patients reaching HbA1c < 7%
* Percentage of patients reaching HbA1c < 6.5%
* Fasting Plasma Glucose (FPG)
* Safety and tolerability

DETAILED DESCRIPTION:
The study duration for each patient is approximately 27 weeks with 3 periods: 2-week screening period followed by 24-week treatment period where patient is assigned to one of the three arms according to randomization, and 3 days follow-up period with a last call phone visit.

ELIGIBILITY:
Inclusion criteria

* Patients with type 2 diabetes mellitus, as defined by the World Health Organization (WHO), diagnosed within one year prior to the screening visit
* Signed informed consent, obtained prior to any study procedure

Exclusion criteria

* Age < 18 and => 78 years old
* HbA1c < 7.6% or > 9%
* BMI > 35 kg/m2
* Diabetes other than type 2 diabetes (e.g.: type 1 diabetes, diabetes secondary to pancreatic disorders, drug or chemical agent intake...)
* Subjects currently receiving or who have received any hypoglycemic agent within 3 months before screening visit

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to week 24

SECONDARY OUTCOMES:
Percentage of patients with HbA1c < 7% | at week 24
Percentage of patients with HbA1c < 6.5 % | at week 24
Change in Fasting Plasma Glucose (FPG) | from baseline week 24
Number of patients reporting adverse events | overt the 24-weeks treatment period
Frequence and incidence of hypoglycemia | over the 24-weeks treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (55):
- Algeria (3):
  - Investigational Site Number 01206, Algeries
  - Investigational Site Number 01203, Oran
  - Investigational Site Number 01205, Sétif
- Colombia (2):
  - Investigational Site Number 17003, El Espinal
  - Investigational Site Number 170001, Manizales
- Egypt (3):
  - Investigational Site Number 81801, Cairo
  - Investigational Site Number 81802, Cairo
  - Investigational Site Number 81803, Cairo
- Guatemala (4):
  - Investigational Site Number 32001, Guatemala City
  - Investigational Site Number 32002, Guatemala City
  - Investigational Site Number 32003, Guatemala City
  - Investigational Site Number 32004, Guatemala City
- India (9):
  - Investigational Site Number 356001, Bangalore
  - Investigational Site Number 356002, Bangalore
  - Investigational Site Number 356006, Ernākulam
  - Investigational Site Number 356003, Indore
  - Investigational Site Number 356009, Lucknow
  - Investigational Site Number 356010, Mumbai
  - Investigational Site Number 356007, Nashik
  - Investigational Site Number 356008, Pune
  - Investigational Site Number 356005, Varanasi
- Iran (3):
  - Investigational Site Number 364001, Tehran
  - Investigational Site Number 364002, Tehran
  - Investigational Site Number 36403, Tehran
- Lebanon (4):
  - Investigational Site Number 42201, Beirut
  - Investigational Site Number 42202, Beirut
  - Investigational Site Number 42203, Chouf
  - Investigational Site Number 422004, Hazmiyeh
- Mexico (2):
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484003, Guadalajara
- Russia (3):
  - Investigational Site Number 643003, Moscow
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643002, Saratov
- South Africa (2):
  - Investigational Site Number 710-002, Durban
  - Investigational Site Number 710-001, Durban
- Tunisia (7):
  - Investigational Site Number 78803, La Marsa
  - Investigational Site Number 78804, La Marsa
  - Investigational Site Number 78805, Sfax
  - Investigational Site Number 78801, Tunis
  - Investigational Site Number 78802, Tunis
  - Investigational Site Number 78806, Tunis
  - Investigational Site Number 78807, Tunis
- Turkey (Türkiye) (6):
  - Investigational Site Number 792-004, Adana
  - Investigational Site Number 792-003, Antalya
  - Investigational Site Number 792-001, Istanbul
  - Investigational Site Number 792-006, Istanbul
  - Investigational Site Number 792-002, Kütahya
  - Investigational Site Number 792-005, Sivas
- Ukraine (3):
  - Investigational Site Number 804001, Kyiv
  - Investigational Site Number 804002, Kyiv
  - Investigational Site Number 804003, Zaporizhzhya
- United Arab Emirates (4):
  - Investigational Site Number 784-001, Dubai
  - Investigational Site Number 784-002, Dubai
  - Investigational Site Number 784-003, Dubai
  - Investigational Site Number 784-004, Sharjah city